CLINICAL TRIAL: NCT03334890
Title: Colorectal Cancer Post-surgical Therapeutic Effect Assessment and Recurrence Monitoring by Methylated SEPT9
Brief Title: CRC Post-surgical Assessment and Recurrence Monitoring
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BioChain (Beijing) Science and Technology, Inc. (Industry)
Collaborators: Chinese PLA General Hospital (Other); First Hospitals affiliated to the China PLA General Hospital (Other Government); 309th Hospital of Chinese People's Liberation Army (Other); Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, LELE SONG, Principal Investigator, 309th Hospital of Chinese People's Liberation Army
Other Study IDs: SEPTMON
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; septin 9; SEPT9; methylation; CEA
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma samples from CRC patients before surgery, one day and seven days after surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: plasma mSEPT9 level — the plasma level of methylated SEPT9

SUMMARY:
The surgical therapeutic effect of stage II-IV CRC patients will be assessed by the plasma mSEPT9 assay, and patients will be followed up by the same assay for recurrence monitoring.

DETAILED DESCRIPTION:
Assessment of surgical therapeutic effect of colorectal cancer (CRC) relies on computer tomography (CT) and serum CEA test. CT cannot be used frequently to monitor the instant change of lesions, while CEA cannot cover all patients due to its low sensitivity. The objective of this study is to assess the performance of the methylated SEPT9 (mSEPT9) in assessing the surgical therapeutic effect of CRC.

This study plans to recruit 50 CRC patients with stage II-IV CRC. Plasma samples before surgery, one day after surgery and seven days after surgery will be collected from each subject. mSEPT9 level will be measured at 3 months, 6 months, 9 months, 12 months, 18 months after surgery and relevant chemotherapy to monitor the possible recurrence of CRC. The mSEPT9 level will be measured by the Epi proColon 2.0 assay. The serum CEA will be measured parallel at the identical time points.

Primary outcomes include the plasma mSEPT9 levels before surgery, one and seven days after surgery.

Secondary outcomes include the serum CEA levels before surgery, one and seven days after surgery. It also includes the size of cancer for each patients, the ratio of patients with mSEPT9 complete response (CR), partial response(PR), progressive disease (PD) and stable disease (SD).

ELIGIBILITY:
Inclusion Criteria:

* stage II-IV CRC patients planning to perform surgery

Exclusion Criteria:

* stage 0-I CRC patients, patients with history of CRC or other cancers, patients not suitable for surgery, pregnant women, patients younger than 30 or older than 80.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stage II-IV CRC patients planning to performe surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
mSEPT9 level | Jan 1, 2016 to Dec 31, 2017
  the Ct values representing the mSEPT9 level in plasma

SECONDARY OUTCOMES:
CEA level | Jan 1, 2016 to Dec 31, 2017
  the serum CEA level
tumor size | Jan 1, 2016 to Dec 31, 2017
  the maximal diameter of tumor measured with CT images
CR,PR,SD,PD | Jan 1, 2016 to Dec 31, 2017
  complete response, partial response, stable disease, progressive disease

CONTACTS AND LOCATIONS:
Overall Officials: Lele Song, M.D.,Ph.D., Study Director — The Chinese PLA 309th Hospital
Locations (4):
- China (4):
  - The Chinese PLA 302th hospital, Beijing
  - The Chinese PLA 309th hospital, Beijing
  - The Chinese PLA general hospital, Beijing
  - The first affiliated hospital of the Chinese PLA general hospital, Beijing

IPD SHARING:
Plan to Share IPD: No